CLINICAL TRIAL: NCT02999997
Title: Randomized Controlled Trial to Evaluate the Rhythm and Music Based Rehabilitation Method the Ronnie Gardiner Method Regarding Dual-task in Individuals With Parkinson's Disease
Brief Title: Evaluation of Ronnie Gardiner Method in Individuals With Parkinson's Disease
Acronym: RGM/PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Petra Pohl, PhD, Researcher, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUH-4865
Record Dates: First submitted 2016-12-10; First posted 2016-12-21 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease
Keywords: Physical therapy modalities; Dual-task performance; Parkinson's disease; Active music therapy; Physical activity
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ronnie Gardiner Method (RGM) (Experimental): Exercising two times/week according to the RGM program in groups of 15 participants (2 groups).
  Interventions: Behavioral: Ronnie Gardiner Method (RGM)
- Control group (No Intervention): Participants in the control group are instructed to live their ordinary life.

INTERVENTIONS:
Behavioral: Ronnie Gardiner Method (RGM) — RGM includes functional exercises consisting of cognitively challenging multi-task exercises. The exercises are performed sitting down or standing up with weight shifting exercises. The practitioner projects unique symbols shaped as red or blue hands and feet on the wall in specific 'choreoscores' of 2-8 bars. Red symbolizes left side of the body, blue the right side. Each symbol is accompanied with a certain movement and sound code. To the sound of rhythmical music the participants follow the symbols beat by beat, performing the movements and pronouncing the word. The exercises are progressed by increasing the tempo of the music, or by using more symbols. The practitioner uses a shirt with the color red on one side, and blue on the other side, in order to facilitate for the participants.
  Other Names: In Sweden and Israel known as RGRM
  Arms: Ronnie Gardiner Method (RGM)

SUMMARY:
Parkinson's disease (PD) is typically associated with cognitive and movement related functional disabilities. One commonly described cognitive complaint is the ability to do several things simultaneously, defined as dual or multiple tasking. The Ronnie Gardiner Method (RGM) is a rhythm and music based rehabilitation intervention that includes components that will train this ability specifically in addition to postural control, motor learning, movement ability and general cognitive function. The aim with the present randomized controlled single-blinded trial is to evaluate the RGM with main focus on dual-task performance, compared to a control group, in individuals with PD. The control group will continue with everyday activities, including ordinary exercise activities, with no additional activity. Both groups will be evaluated pre-, post-, and after 3 months post intervention. Following outcome measures will be analyzed:

1. dual task performance (motor-motor, and motor-cognitive)
2. level of physical activity, motor function and balance
3. cognitive function including memory and spatial function
4. health-related quality of life, fear of falling, and freezing of gait
5. qualitative interviews from focus group discussions

DETAILED DESCRIPTION:
Patients with Parkinson's disease at the neurological department of University Hospital of Linköping are included and randomized to either the rhythm and music based rehabilitation method Ronnie Gardiner Method or to a control group with no other activity other than everyday activities including habitual exercise. Timed Up and Go (TUG) cognitive and TUG manual will be used to evaluate dual-task performance. The intervention will take place twice weekly for twelve weeks in a neurological rehabilitation facility, and will be led by a highly skilled physiotherapist with ten years of practice from the Ronnie Gardiner Method.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease, stage 1,5 to 4 on the Hoehn & Yahr scale, community dwelling, stable medication, being able to walk at least 10 meters, being able to transport to the intervention facility, being able to follow instructions in Swedish

Exclusion Criteria:

* parkinsonism of other origin, color blindness, severely impaired vision or hearing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Cognitive (TUGcog) (motor-cognitive dual task) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Time in seconds to complete the following sequence: stand up from a chair, walk 3 meters, turn, walk back to the chair and sit down with the addition of counting backwards with 7 from 100, 90, 80, 70, 60, or 50. Number of errors are noted. Higher speed indicated better function.
Timed Up and Go manual (TUG manual) (motor-motor dual task) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Time in seconds to complete the following sequence: stand up from a chair, walk 3 meters, turn, walk back to the chair and sit down with the additional task to carry a tray with two glasses of water. Higher speed indicates better function.

SECONDARY OUTCOMES:
Dual-task cost (DTC) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Measuring the difference between Timed Up and Go (TUG) single task and TUG cognitive and manual respectively
Mini-BESTest (Balance Evaluation Systems Test) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  A balance test focusing on dynamic balance and can be conducted in 10-15 minutes.
Four Step Square Test, FSST | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Patient steps over four canes set-up like a cross on the floor with the tips of the canes facing together. At the start of the test, the patient stands on the upper left square (in Square 1, facing Square 2). The stepping sequence is (clockwise): Square 1, Square 2, Square 4, Square 3, return to Square 1 with the feet. Then (counterclockwise): Back to Square 3, Square 4, Square 2, and end in Square 1 with both feet.
Berg Balance Scale | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Static and dynamic activities of varying difficulty are performed. Item-level scores range from 0-4, determined by ability to perform the assessed activity. Item scores are summed. Maximum score = 56
Chair stand 30 seconds | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Standing up and sitting down, hands crossed over chest, as many times as possible for 30 seconds.
Montreal Cognitive Assessment (MoCA) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Screening of cognitive function. License has been approved.
Auditory memory test, direct and delayed | Change from Baseline through study completion (at 12 weeks) and at 3 months
  A text is read to the patient. The patient is then required to reproduce the text as exactly as possible, and then again after appr. 10 minutes.
Symbol Digit Modalities Test (SDMT) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  A code key is presented to the patient where each code key represents a number between 1 and 9. The patient is then required to solve as many codes as possible in 90 seconds.
Victoria Stroop test | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Colored words are presented to the patient but in a different color than the word says, eg. the word BLUE appears in the color red and the patient is required to say "red", and not read the word "blue".
Grooved Pegboard | Change from Baseline through study completion (at 12 weeks) and at 3 months
  The patient is required to move a number of metal sticks from one side to another as fast as possible. A measure of fine motor control.
Trail Making Test A and B | Change from Baseline through study completion (at 12 weeks) and at 3 months
  The patient is required to draw a line between the numbers 1 to 25 (A), and between the numbers 1 to 13 and vary to the letters A to L, i.e. 1-A-2-B-3-C, etc, without lifting the pen from the paper.
Rey complex figure | Change from Baseline through study completion (at 12 weeks) and at 3 months
  The patient is required to copy a figure twice: the first time from a model in front of him/her; the second time without the model by memory only.
WHODAS 2.0 | Baseline
  A questionnaire based on the International Classification of Functioning (ICF) for assessing impairments and function.
Freezing of gait questionnaire | Change from Baseline through study completion (at 12 weeks) and at 3 months
  A questionnaire with questions about freezing of gait
Parkinson's disease questionnaire 39 items (PDQ-39) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  A questionnaire for quality of life in people with Parkinson's disease. License as been approved.
Falls Efficacy Scale International (FES-I) | Change from Baseline through study completion (at 12 weeks) and at 3 months
  A questionnaire related to fear of falling.
Actigraphy with GeneActiv Armband | Change from Baseline through study completion (at 12 weeks) and at 3 months
  Actigraphy is a method to evaluate physical activity in a research person´s normal life. GeneActiv is used to record number of steps daily but also time spent lying and standing which will give information about the activity.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Pohl, PhD, RPT, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- Neurological clinic, Linkoeping Universityhospital, Linköping, Östergötland County, Sweden

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886